CLINICAL TRIAL: NCT03341975
Title: Enhanced SexHealth Intervention to Improve Adolescent Outcomes: A Clinical Trial
Brief Title: Enhanced SexHealth Intervention to Improve Adolescent Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17010079
Record Dates: First submitted 2017-11-06; First posted 2017-11-14 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Sexually Transmitted Diseases; Reproductive Behavior
MeSH Terms: conditions — Sexually Transmitted Diseases; Reproductive Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): They will receive the same pamphlet as controls and the enhanced ED SexHealth intervention with the educator. Based on behaviors, CDS system recommendations (generated from screening survey responses only for intervention participants), and discussions, participants may be offered testing (for pregnancy, gonorrhea/chlamydia, and /or HIV), hormonal birth control, condoms, emergency contraception (for immediate or future use), treatment for previously diagnosed (yet untreated) infection with gonorrhea/chlamydia, and a scheduled appointment at Adolescent Clinic (for ongoing care, including repeat STI/HIV testing if needed). All services will be provided at point of care, costs will be covered by the study.
  Interventions: Behavioral: SexHealth
- Control (No Intervention): They will receive a printed health pamphlet and a list of local resources with the phone number for Adolescent Clinic. Participants will then be referred back to their ED provider, who will provide their standard care.

INTERVENTIONS:
Behavioral: SexHealth — To enhance and test our ED SexHealth intervention that provides risk reduction counseling and point-of-care services as well as connections to sustainable, non-episodic sources of care.
  Arms: Intervention

SUMMARY:
This is an adaptive trial with an initial Formative Revision Process followed by a Randomized Controlled Trial (RCT). Up to 500 adolescents will be consented into this study to achieve 6 completed subjects for the formative process and 86 completed subjects for the RCT.

DETAILED DESCRIPTION:
In a randomized controlled trial at a pediatric emergency department, sexually active adolescents will receive the control (i.e., printed materials) or intervention (i.e., motivationally-guided facilitation) arm delivered by a health educator. The tablet-based, interactive intervention includes motivational techniques to promote risk reduction, condom skills training, and tailored service recommendations. The primary outcome is uptake of ≥1 service at the index visit (i.e., counseling, condoms, emergency contraception for immediate or future use, pregnancy/sexually transmitted infection (STI)/HIV testing, STI treatment, and clinic referral). We assess feasibility (i.e., intervention completion, recommendations discussed, and satisfaction). Participants report sexual risk and care-seeking behaviors at 2, 4, and 6 months. We compare uptake between arms using Fisher exact tests.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14-19 years old
* Reside within 30 minutes travel time
* Report previous sexual activity

Exclusion Criteria:

* Subjects who are unable to provide consent (i.e., determined to be too ill by the ED team, have cognitive impairment due to chronic condition or acute medical concern)
* Subjects in police custody
* Subjects seeking care due to sexual assault or psychiatric emergency
* Subjects who do not speak English
* Subjects who are patients under the clinical care of a study investigator working in the ED

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Miller, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Miller MK, Catley D, Adams A, Staggs VS, Dowd MD, Stancil SL, Miller E, Satterwhite CL, Bauermeister J, Goggin K. Brief Motivational Intervention to Improve Adolescent Sexual Health Service Uptake: A Pilot Randomized Controlled Trial in the Emergency Department. J Pediatr. 2021 Oct;237:250-257.e2. doi: 10.1016/j.jpeds.2021.06.007. Epub 2021 Jun 16. PMID 34144031

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 44 | 47
Completed | 44 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 44 | 47 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.8 (0.7) | 17.0 (0.8) | 16.9 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 34 | 65
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 11 | 18
  Not Hispanic or Latino | 37 | 36 | 73
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 30 | 58
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 44 | 47 | 91
Commercial Insurance [Count of Participants; unit: Participants] | 8 | 9 | 17
Genitourinary complaint [Count of Participants; unit: Participants] | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Uptake of 1 or More Health Services
Description: Any 1 or more of the following services: Testing for pregnancy, gonorrhea/chlamydia, and/or HIV, hormonal birth control, condoms, emergency contraception (for immediate or future use), treatment for previously diagnosed (yet untreated) infection with gonorrhea/chlamydia, appointment for clinic referral.
Time Frame: Index visit
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 44 | 47
Participants | 43 | 33

ADVERSE EVENTS:
Time Frame: Information was collected at index visit and at six month follow-up.
Description: Information was collected at index visit and at six month follow-up.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/47
Other Adverse Events (participants affected / at risk) | 0/44 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT03341975/Prot_SAP_000.pdf